CLINICAL TRIAL: NCT06460909
Title: Randomised Study Evaluating the Interest of Psychological Support of Patients Waiting for Hallux Valgus Surgery
Acronym: PrePS HV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP220331; 2022-A00381-42 (Registry Identifier: IDRCB)
Record Dates: First submitted 2024-05-30; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-05

CONDITIONS: Hallux Valgus Surgery
Keywords: Hallux Valgus Surgery; Psychological Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychological support arm (Experimental): Patients randomized with psychological intervention.
  Interventions: Other: Psychological support
- Without support (No Intervention): Patients with routine care with psychological support.

INTERVENTIONS:
Other: Psychological support — An interview with the psychologist before surgery.
  Arms: Psychological support arm

SUMMARY:
Catastrophizing is a negative evaluation of events. What surgery concerns, pain catastrophizing is one of the main risks of postoperative pain and / or poor functional recovery. The best survey to evaluate pain catastrophizing is the PCS (Pain Catastrophizing Scale). According to the authors, catastrophizers report more negative pain related thoughts, more emotional distress and more pain than non-catastrophizers. The PCS is a significant predictor of pain intensity and so of poor functional recovery.

It is already well known that anxiety and catastrophizing predict postoperative pain.

The actual studies focus mainly on functional recovery of knee and hip arthroplasties, but less on pain and functional recovery of hallux valgus surgery.

According to several authors, adapted psychological support of preoperative catastrophizing could allow a better postoperative evolution.

Our hypothesis is that a preoperative psychological consultation of catastrophizing patients is efficient to lower pain catastrophizing in adult patients undergoing a surgical operation for hallux valgus.

The first objective is to evaluate the impact of a psychological support of preoperative pain catastrophizing during a hallux valgus surgery.The principal evaluation scale is the pain catastrophizing score before and after surgery.

The second objective is to evaluate the pain and functional recovery of pain catastrophizing patients. The criteria of this survey are: anxiety score (usual and actual), pain and function according to the FAOS (Foot and Ankle Outcome Score) pain (Analogic Visual Scale).

ELIGIBILITY:
Inclusion Criteria:

* Adult over 18
* Independent, living in its own home
* Affiliated at a social security
* Consent signed
* Waiting for a Hallux Valgus surgery.

Exclusion Criteria:

* Not Able to understand french language
* Patient refusal
* Under guardianship
* Under french AME system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2024-11-02 (Estimated); Study Completion 2025-02-02 (Estimated)

PRIMARY OUTCOMES:
Impact of preoperative psychological support on pain catastrophizing | at baseline
  By State portion of the Spielberger State-Trait Anxiety Inventory STAI.

SECONDARY OUTCOMES:
Pain evaluate of catastrophizing patients | at baseline
  By American Orthopaedic Foot and Ankle Society (AOFAS).

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Hélène Sandiford, Principal Investigator — Ambroise Paré hospital - APHP
Locations (1):
- Orthopedia and traumatological department, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: Undecided